CLINICAL TRIAL: NCT00274729
Title: MUFObes: MonoUnsaturated Fatty Acids in Obesity - a Comparison Between 3 Different Diets in Weight Maintenance and the Prevention of Lifestyle Diseases in Obese Subjects. A Randomised, Long-term Intervention Study.
Brief Title: Mono Unsaturated Fatty Acids in Obesity - Weight Maintenance and Prevention of Lifestyle Diseases in Obese Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Aarhus University Hospital (Other); University Hospital, Gentofte, Copenhagen (Other); Rigshospitalet, Denmark (Other); Technical University of Denmark (Other); Harvard School of Public Health (HSPH) (Other); Boston Children's Hospital (Other); Danish Meat Research Institute (Other); Danisco (Industry); The Danish Dairy Research Foundation, Denmark (Other); Various FOOD sponsors have provided groceries for the dietary intervention (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KF 01-172/03
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2006-01

CONDITIONS: Overweight; Obesity
Keywords: Dietary intervention; High-carbohydrate diet; High-fat diet; Moderate-fat diet; Obesity; Weight maintenance; Body composition; Glucose metabolism; Cardiovascular disease; Appetite regulation; Energy expenditure
MeSH Terms: conditions — Overweight; Obesity; Cardiovascular Diseases | interventions — Adiposity

INTERVENTIONS:
Behavioral: Mono Unsaturated Fatty Acids in Obesity

SUMMARY:
The purpose of this study is to investigate the effect of three diets different in type and amount of fat in weight maintenance and prevention of life-style diseases in obese subjects.

DETAILED DESCRIPTION:
The obesity epidemic has raised concerns, because of complications such as type 2 diabetes, cardiovascular disease and certain types of cancer. Much conflict and confusion about the optimal diet for weight control exists among the public.

The current dietary recommendations aim at reducing the total fat in the diet to less than 30% of calories, increasing carbohydrates to 55-60%, and protein from lean meat and dairy products to 15-20%, and to keep the intake of sugar sweetened soft-drinks limited. There is good evidence from meta-analyses of intervention studies that a low fat diet can prevent weight gain in normal weight individuals, induce a small but clinically relevant weight loss in overweight individuals, and also reduce the risk of cardiovascular disease and type 2 diabetes.

However this recommended diet may not be of the optimal composition in preventing the progressive increase in obesity and lifestyle diseases. The traditional dietary recommendation has been challenged by the epidemiologist Walter Willett, Harvard Medical School in Boston. He claims that dietary fat is less important for the development of obesity, and that the fat content of the diet can be 40-45% of the energy providing from mainly mono- and polyunsaturated fatty acids. Based on mainly large-scale observational studies ('Nurses Health Study') he has developed new dietary guidelines, expressed as a new diet pyramid. In contrast to the current guidelines, more plant oils and plant foods, limited animal products, such as meat and dairy products (even lean products), and increased intake of olive oil, nuts, etc., e.g. guidelines closer to the "Mediterranean Diet".

There is circumstantial evidence to support that this moderate fat, MUFA-rich diet will have a beneficial effect on some of the traditional risk factors for cardiovascular disease and type-2 diabetes. However, there is also growing concern that the increased total fat content will lead to weight gain and increased risk of obesity, and secondary to this, type-2 diabetes and cardiovascular disease. This debate has now been taken up by some of the finest scientific journals. To test this hypothesis the largest and longest dietary intervention trial in Denmark is carried out at the Department of Human Nutrition.

The objective is to identify the diet and diet components most effective for protection against weight gain, weight regain and prevention of life-style diseases in obese subjects. The three diets tested are according to:

1. Willetts new dietary recommendations. High in mono unsaturated fat and low in glycemic index (50 subjects).
2. The traditional dietary recommendations. Low in fat and medium in glycemic index (50 subjects).
3. The average Danish diet (Control). High in fat and high in glycemic index (25 subjects).

The diets are ad libitum (i.e. no restriction in calorie intake), but very strict in dietary composition.

ELIGIBILITY:
Inclusion Criteria:

* Age: 16-35 years
* Body mass index (kg/m2): 28-36

Exclusion Criteria:

* Body weight fluctuations > 3 kg over the previous 2 months
* Smoking

Presence of:

* Cardiovascular diseases, cancer tumours, kidney or lever diseases, infections or endocrinological diseases, malabsorption disorders
* Systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg
* Hypercholesterolemia with changes in pharmacological treatment within the last 2 months
* Regular use of medicine other than birth pills, any psychological disorders, known or presumed abuse of alcohol, allergies to any food, special diets (eg. vegetarian) or particular dislikes
* Pregnancy, lactating or planning pregnancy within 18 month from enrolment

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 125
Dates: Start 2004-01; Study Completion 2008-06

PRIMARY OUTCOMES:
Changes in body weight
Weight loss maintenance efficacy (>5% and >10%)
Body composition (whole body DEXA-scanning)
Drop-out rate
Glucose metabolism (Oral Glucose Tolerance Test)
Endothelium function (flow-mediated vasodilatation, FMD)

SECONDARY OUTCOMES:
Changes in:
Blood lipids
Blood glucose
HbA1c
Insulin
Blood coagulation factors
Waist
Waist/hip-ratio
Blood pressure
Appetite & diet palatability
Appetite regulating hormones (during meal test)
Visual analogue scale (VAS) (during meal test)
Energy expenditure (24 hour whole body indirect calorimetry)

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, MD DMSC, Principal Investigator — Department of Human Nutrition, The Royal Veterinary & Agricultural University

REFERENCES:
- [Derived] Hjorth MF, Due A, Larsen TM, Astrup A. Pretreatment Fasting Plasma Glucose Modifies Dietary Weight Loss Maintenance Success: Results from a Stratified RCT. Obesity (Silver Spring). 2017 Dec;25(12):2045-2048. doi: 10.1002/oby.22004. Epub 2017 Oct 6. PMID 28985039
- [Derived] Due A, Larsen TM, Mu H, Hermansen K, Stender S, Astrup A. Comparison of 3 ad libitum diets for weight-loss maintenance, risk of cardiovascular disease, and diabetes: a 6-mo randomized, controlled trial. Am J Clin Nutr. 2008 Nov;88(5):1232-41. doi: 10.3945/ajcn.2007.25695. PMID 18996857
- [Derived] Due A, Larsen TM, Hermansen K, Stender S, Holst JJ, Toubro S, Martinussen T, Astrup A. Comparison of the effects on insulin resistance and glucose tolerance of 6-mo high-monounsaturated-fat, low-fat, and control diets. Am J Clin Nutr. 2008 Apr;87(4):855-62. doi: 10.1093/ajcn/87.4.855. PMID 18400707